CLINICAL TRIAL: NCT01449877
Title: Influence of Trimethoprim-sulfamethoxazole for the Recurrence of Retinochoroiditis Toxoplasma Gondii
Brief Title: Influence of Trimethoprim-Sulfamethoxazole for the Recurrence of Ocular Toxoplasmosis
Acronym: ISROT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Joao Paulo Felix, MD, University of Campinas, Brazil
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 356591
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Ocular Toxoplasmosis
Keywords: Ocular Toxoplasmosis; Retinochoroiditis; Prophylaxis
MeSH Terms: conditions — Toxoplasmosis, Ocular; Chorioretinitis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Sulfamethoxazole; Trimethoprim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trimethoprim-Sulfamethoxazole (Active Comparator): 1 tablet every other day, morning.
  Interventions: Drug: Trimethoprim-Sulfamethoxazole
- Starch tablet (Placebo Comparator): 1 starch tablet every other day, morning.
  Interventions: Drug: Trimethoprim-Sulfamethoxazole

INTERVENTIONS:
Drug: Trimethoprim-Sulfamethoxazole — Sulfamethoxazole 800mg + Trimethoprim 160mg / tablet. In treatment of acute phase, 1 tablet 12/12h 45 days. After acute phase, 1 tablet every other day, morning, 311 days. Placebo tablet - Composition: starch. After acute phase, 1 tablet every other day, morning, 311 days.
  Other Names: Sulfamethoxazole 800mg + Trimethoprim 160mg = Bactrim F.

SUMMARY:
The investigators study aims to determine the effect of prophylactic therapy with Trimethoprim-sulfamethoxazole on the recurrences of toxoplasma retinochoroiditis gondii. This is a randomized, double-masked, in patients with eye condition of acute Toxoplasma gondii retinochoroiditis. Volunteers will be recruited with a previous diagnosis of chorioretinitis presumed Toxoplasma gondii, which show active lesions compatible with recurrence. After the acute phase of treatment of all patients [1 tablet Trimethoprim-sulfamethoxazole (800/160mg) 12/12h during 45 days], the same Stratified by gender) will be randomized in a 1:1 ratio between the group 1 - TMP-SMZ (prophylactic treatment with trimethoprim-sulfamethoxazole 1 tablet every other day for 311 days) or group 2 - placebo (consisting of a placebo pill containing no active ingredient of similar appearance to trimethoprim-sulfamethoxazole, 1 tablet every other day for 311 days). The primary outcomes are incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 12, 36, 48, 60, 72, 84, 96, 108, and 120 months. Patients will be followed during the ten years in uveitis clinic at intervals defined as follows: return weekly for 4 weeks, then monthly for 2 months, then each 3 months for 9 months, and finally annually for 10 years.

DETAILED DESCRIPTION:
The protozoan Toxoplasma gondii is an obligate intracellular parasite, a common cause of intraocular inflammation in the world. The treatment of toxoplasmosis is the sulfonamide group of drugs, which acts on tachyzoites forms, no acting on bradyzoites, that grown from latent focus located on boards and are responsible for recurrence. The investigators study aims to determine the effect of prophylactic therapy with Trimethoprim-sulfamethoxazole on the recurrences of toxoplasma retinochoroiditis gondii. This is a randomized, double-masked, in patients with eye condition of acute Toxoplasma gondii retinochoroiditis. The study population consists of patients treated at Ophthalmology department, University of Campinas. They present symptoms compatible with a diagnosis of recurrent ocular toxoplasmosis. Volunteers will be recruited with a previous diagnosis of chorioretinitis presumed Toxoplasma gondii, which show active lesions compatible with recurrence. After the acute phase of treatment of all patients [1 tablet Trimethoprim-sulfamethoxazole (800/160mg) 12/12h during 45 days], the same Stratified by gender) will be randomized in a 1:1 ratio between the group 1 - TMP-SMZ (prophylactic treatment with trimethoprim-sulfamethoxazole 1 tablet every other day for 311 days) or group 2 - placebo (consisting of a placebo pill containing no active ingredient of similar appearance to trimethoprim-sulfamethoxazole, 1 tablet every other day for 311 days). The definition of a patient with recurrent episode of chorioretinitis Toxoplasmosis is the presence of old scars of chorioretinitis, associated with satellite active lesions chorioretinitis with positive IgG for toxoplasmosis. The new recurrence was treated with 1 tablet Trimethoprim-sulfamethoxazole (800/160mg) 12/12h during 45 days. The patients will be tested for visual acuity, examination biomicroscopy, tonometry, fundus photography and indirect ophthalmoscopy. In each study, patients will be randomized in blocks of four (two in group I and two Group II) with stratification by gender. The primary outcomes are incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 12, 36, 48, 60, 72, 84, 96, 108, and 120 months. It was planned a minimum sample of 140 patients (70 in group I and 70 in group II). Assuming an incidence of 6% recurrence in group A, this sample will have a 80% power to detect a difference of 18% between groups. The results of this analysis will be considered significant if p <0.05. The main variables are age, sex, presence of unilateral or bilateral eye injury, number of recurrences, number and location of lesions, and previous treatment for ocular toxoplasmosis. Patients will be followed during the ten years in uveitis clinic at intervals defined as follows: return weekly for 4 weeks, then monthly for 2 months, then each 3 months for 9 months, and finally annually for 10 years. Patients will be trained to return immediately if they have any of the following symptoms: decreased visual acuity, photophobia, floaters or ocular hyperemia. Adverse events will be monitored. The definition of a patient with a recurrent episode of chorioretinitis Toxoplasmosis is the presence of old scars of chorioretinitis, associated with active satellite lesions chorioretinitis with positive IgG for toxoplasmosis. To data collection, will be used semi-structured questionnaire, containing the patient record, age, gender, visual acuity by ETDRS chart, the affected eye and previous treatment for ocular toxoplasmosis.

ELIGIBILITY:
Inclusion Criteria:

* Positive IgG result for toxoplasmosis (IgG)
* Ipsilateral scars of retina compatible with previous episode of toxoplasmosis retinochoroiditis
* Unilateral active lesion of chorioretinitis

Exclusion Criteria:

* Under 18 years of age
* Immunosuppressed patients
* Use of immunosuppressive treatments
* Concomitant chorioretinitis of other causes
* Pregnancy
* Allergy to Sulfonamides

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 12 months. | One year
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 36 months. | Three years
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 48 months. | Four years
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 60 months. | Five years
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 72 months. | Six years
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 84 months. | Seven years
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 96 months. | Eight years
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 108 months. | Nine years
Incidence of episodes of recurrent chorioretinitis by toxoplasmosis in the follow up of 120 months. | Ten years

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo PC Lira, PhD, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas - Ophthalmology Department, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Opremcak EM, Scales DK, Sharpe MR. Trimethoprim-sulfamethoxazole therapy for ocular toxoplasmosis. Ophthalmology. 1992 Jun;99(6):920-5. doi: 10.1016/s0161-6420(92)31873-1. PMID 1630782
- [Background] Soheilian M, Sadoughi MM, Ghajarnia M, Dehghan MH, Yazdani S, Behboudi H, Anisian A, Peyman GA. Prospective randomized trial of trimethoprim/sulfamethoxazole versus pyrimethamine and sulfadiazine in the treatment of ocular toxoplasmosis. Ophthalmology. 2005 Nov;112(11):1876-82. doi: 10.1016/j.ophtha.2005.05.025. Epub 2005 Sep 19. PMID 16171866
- [Background] Gilbert RE, See SE, Jones LV, Stanford MS. Antibiotics versus control for toxoplasma retinochoroiditis. Cochrane Database Syst Rev. 2002;(1):CD002218. doi: 10.1002/14651858.CD002218. PMID 11869630
- [Result] Silveira C, Belfort R Jr, Muccioli C, Holland GN, Victora CG, Horta BL, Yu F, Nussenblatt RB. The effect of long-term intermittent trimethoprim/sulfamethoxazole treatment on recurrences of toxoplasmic retinochoroiditis. Am J Ophthalmol. 2002 Jul;134(1):41-6. doi: 10.1016/s0002-9394(02)01527-1. PMID 12095806
- See also: University of Campinas — http://www.fcm.unicamp.br